CLINICAL TRIAL: NCT00302068
Title: Understanding the Prognostic Benefits of Exercise and Anti-depressant Therapy (UPBEAT)
Brief Title: Exercise to Treat Depression in Individuals With Coronary Heart Disease
Acronym: UPBEAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00011980; R01HL080664-01A1 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-05

CONDITIONS: Depression; Heart Diseases
Keywords: Exercise
MeSH Terms: conditions — Depression; Heart Diseases; Motor Activity | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Supervised aerobic exercise, three times per week for 16 weeks.
  Interventions: Behavioral: Supervised Aerobic Exercise
- 2 (Active Comparator): Sertraline (Zoloft), for 16 weeks.
  Interventions: Drug: Sertraline
- 3 (Placebo Comparator): Placebo control, for 16 weeks.
  Interventions: Drug: Placebo Pill.

INTERVENTIONS:
Behavioral: Supervised Aerobic Exercise — Supervised aerobic exercise, three times per week, for 16 weeks.
  Arms: 1
Drug: Sertraline — Sertraline (Zoloft), daily, for 16 weeks.
  Arms: 2
Drug: Placebo Pill. — Placebo pill, daily, for 16 weeks.
  Arms: 3

SUMMARY:
Some individuals with coronary heart disease (CHD) suffer from depression and use antidepressant medications to reduce symptoms. However, preliminary research has shown that exercise may be a more effective way to treat depression in these individuals. The purpose of this study is to evaluate the effects of exercise in reducing depression and improving heart function in individuals with CHD.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is caused by a narrowing of the small blood vessels that supply blood and oxygen to the heart. It is the leading cause of death in the United States. Recent evidence has suggested that depression is a significant risk factor for individuals with CHD and may place additional strain on the heart. Selective serotonin reuptake inhibitors (SSRIs), a type of antidepressant medication, have been shown to be especially effective at reducing depression symptoms, particularly for individuals with CHD. However, many people fail to benefit from medication alone or they experience negative side effects. Therefore, a need exists to identify alternative approaches for treating depression in individuals with CHD. Preliminary research has shown that exercise may be an effective way to improve mood and treat depression. More research, however, is needed to confirm the benefits of exercise in individuals with CHD. The purpose of this study is to compare the effectiveness of a supervised exercise program, antidepressant treatment, and placebo in reducing depression and improving heart function in individuals with CHD.

This 16-week study will enroll adults with a history of CHD and depression. Participants will be randomly assigned to an aerobic exercise program, antidepressant medication, or placebo. At study entry, standardized psychological questionnaires will be completed and depression levels and exercise tolerance will be assessed. Participants' heart function will be evaluated through measures of flow-mediated vasodilatation, inflammation, platelet function, baroreflex, and heart rate variability. Participants assigned to the exercise program will be required to engage in structured aerobic exercise. Participants assigned to antidepressant medication will receive sertraline, an SSRI or placebo. The treating psychiatrist will be blinded to pill condition and will use supportive measures to help manage medication side effects. Outcome assessors will be unaware of patients' treatment assignments, and only the research pharmacist will be aware of which patients are assigned to sertraline or to placebo.

At Week 16, participants will return to the clinic for repeat assessments of baseline measures. A follow-up evaluation will occur six months following the end of treatment, and participants' depression levels and clinical status will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Persistent depressive symptoms that may include the following: depressed mood; diminished interest or pleasure in activities; change in appetite; insomnia or hypersomnia; psychomotor agitation or retardation; fatigue or loss of energy; feelings of worthlessness or inappropriate guilt; diminished ability to think or concentrate; or recurrent thoughts of death or suicidal ideations
* Documented history of coronary heart disease (i.e., a prior heart attack, coronary artery bypass graft, or greater than 75% stenosis in at least one coronary artery)

Exclusion Criteria:

* Experienced an acute heart attack or any revascularization procedure (i.e., CABG or percutaneous transluminal coronary angioplasty) within 60 days of study entry
* Left ventricular ejection fraction <30% with labile ECG changes prior to testing
* Currently using a pacemaker
* Resting blood pressure greater than 160/100 mmHg
* Left main disease >50%
* Failure to meet our criteria for depression or achieve a score of ≥9 on the Beck Depression Inventory-II
* Any other concurrent psychiatric intervention
* Primary psychiatric diagnosis other than Major or Minor Depressive Episode
* Primary diagnosis of the following psychiatric disorders: schizophrenia, bipolar disorder, schizoaffective disorder, other psychotic disorder, dementia, current delirium, current obsessive compulsive disorder
* Experienced psychotic symptoms during the current depressive episode
* Current abuse or dependence on alcohol or other drugs
* Acute suicide risk
* Patients who, during the course of the study, would likely require treatment with additional psychotherapeutic agents
* Significant medical conditions that would make exercise or sertraline use medically inadvisable (e.g., unstable angina, heart attack within the 3 months prior to study entry, musculoskeletal problems, or congestive heart failure)
* Abnormal thyroid-stimulating hormone (TSH) level and glucose level greater than or equal to 126 mg/dL
* Patients who would not be able to be randomized to either the drug (e.g., adverse cardiac events such as prolonged QT interval, allergic responses) or exercise (e.g., musculoskeletal problems, abnormal cardiac response to exercise, such as exercise-induced VT, abnormal blood pressure response, etc.)
* Currently using medications that would make exercise or sertraline use medically inadvisable (e.g., clonidine, dicumarol, warfarin, anticonvulsants, or MAO inhibitors)
* Current uncontrolled medical condition that could be causing the depressive symptoms (e.g., thyroid dysfunction, anemia)
* Pregnant, planning to get pregnant during the study period, or lactating
* Herbal supplements with purported mood effects (e.g., St. John's wort, valerian, gingko)
* Current use of antidepressant medication
* Currently participating in psychotherapy
* Currently participating in regular aerobic exercise
* Documented failure to respond to sertraline therapy

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-07; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Blumenthal, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Babyak M, Blumenthal JA, Herman S, Khatri P, Doraiswamy M, Moore K, Craighead WE, Baldewicz TT, Krishnan KR. Exercise treatment for major depression: maintenance of therapeutic benefit at 10 months. Psychosom Med. 2000 Sep-Oct;62(5):633-8. doi: 10.1097/00006842-200009000-00006. PMID 11020092
- [Background] Blumenthal JA, Babyak MA, Moore KA, Craighead WE, Herman S, Khatri P, Waugh R, Napolitano MA, Forman LM, Appelbaum M, Doraiswamy PM, Krishnan KR. Effects of exercise training on older patients with major depression. Arch Intern Med. 1999 Oct 25;159(19):2349-56. doi: 10.1001/archinte.159.19.2349. PMID 10547175
- [Background] Blumenthal JA, Sherwood A, Babyak MA, Watkins LL, Waugh R, Georgiades A, Bacon SL, Hayano J, Coleman RE, Hinderliter A. Effects of exercise and stress management training on markers of cardiovascular risk in patients with ischemic heart disease: a randomized controlled trial. JAMA. 2005 Apr 6;293(13):1626-34. doi: 10.1001/jama.293.13.1626. PMID 15811982
- [Background] Dunn AL, Trivedi MH, Kampert JB, Clark CG, Chambliss HO. Exercise treatment for depression: efficacy and dose response. Am J Prev Med. 2005 Jan;28(1):1-8. doi: 10.1016/j.amepre.2004.09.003. PMID 15626549
- [Background] Dunn AL, Trivedi MH, Kampert JB, Clark CG, Chambliss HO. The DOSE study: a clinical trial to examine efficacy and dose response of exercise as treatment for depression. Control Clin Trials. 2002 Oct;23(5):584-603. doi: 10.1016/s0197-2456(02)00226-x. PMID 12392873
- [Background] Lett HS, Blumenthal JA, Babyak MA, Sherwood A, Strauman T, Robins C, Newman MF. Depression as a risk factor for coronary artery disease: evidence, mechanisms, and treatment. Psychosom Med. 2004 May-Jun;66(3):305-15. doi: 10.1097/01.psy.0000126207.43307.c0. PMID 15184688
- [Background] Blumenthal JA, Sherwood A, Babyak MA, Watkins LL, Smith PJ, Hoffman BM, O'Hayer CV, Mabe S, Johnson J, Doraiswamy PM, Jiang W, Schocken DD, Hinderliter AL. Exercise and pharmacological treatment of depressive symptoms in patients with coronary heart disease: results from the UPBEAT (Understanding the Prognostic Benefits of Exercise and Antidepressant Therapy) study. J Am Coll Cardiol. 2012 Sep 18;60(12):1053-63. doi: 10.1016/j.jacc.2012.04.040. Epub 2012 Aug 1. PMID 22858387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in June 2006 and ended in September 2010. Participants were recruited from physician referrals, community-based screenings, and mass media advertisements.
Groups:
- Supervised Aerobic Exercise: Patients will attend 3 supervised group aerobic exercise sessions per week for 16 weeks. On the basis of peak heart rate achieved during the initial treadmill test, patients are assigned training ranges equivalent to 70% to 85% maximal heart rate reserve. Each aerobic session will consist of 30 min of walking or jogging on a treadmill at an intensity that would maintain heart rate within the assigned training range.
- Sertraline (Zoloft): Participants are given the selective serotonin reuptake inhibitor sertraline. Medications are taken once daily; the dosage depends on the clinical response, but usually, each patient will start at 50 mg (1 pill) of drug and progress up to 200 mg (4 pills), contingent on therapeutic response and the presence of side effects.
- Placebo Control: Participants are given a matching placebo. Medications are taken once daily; the dosage depends on the clinical response, but usually, each patient will start at 50 mg (1 pill) of placebo and progress up to 200 mg (4 pills), contingent on therapeutic response and the presence of side effects.
Period: Overall Study
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Started | 37 | 40 | 24
Completed | 36 | 36 | 23
Not Completed | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control | Total
Number analyzed (Participants) | 37 | 40 | 24 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 14 | 60
  >=65 years | 15 | 16 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (11.0) | 63.4 (10.2) | 63.5 (11.4) | 63.9 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 4 | 32
  Male | 24 | 25 | 20 | 69
Region of Enrollment [Number; unit: participants]
  United States | 37 | 40 | 24 | 101

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale
Description: The Hamilton Depression Rating Scale ranges from 0 to 52, with lower scores reflecting lower levels of depression and higher scores greater severity of depression.
Time Frame: Measured at 16 weeks
Population: All completed subjects plus 1 subject in the sertraline arm who did not complete but provided assessment data.
Measure: Mean (95% Confidence Interval); unit: Raw changes in Ham-D scores
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Number analyzed (Participants) | 36 | 37 | 23
Raw changes in Ham-D scores | -7.5 [-9.8 to -5.0] | -6.1 [-8.4 to -3.9] | -4.5 [-7.6 to -1.5]

2. Secondary Outcome: Heart Rate Variability (HRV)
Description: HRV is the variation in the time interval between heart beats. ECG was recorded for 24 hours on a 3-channel digital compact ash Holter recorder. During the recording period, patients engaged in their normal patterns of activity. ECG data were downloaded and edited using the Pathfinder digital ambulatory ECG analyzer (DelMar Reynolds, lrvine, California) and HRV was estimated from the standard deviation of all normal R-R intervals (SDNN)
Time Frame: Baseline, 16 weeks
Population: Analysis based on 93 participants with valid baseline measurements.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Number analyzed (Participants) | 33 | 38 | 22
millisecond
  Baseline | 116 (36) | 120 (39) | 123 (24)
  16 Weeks | 122 (35) | 118 (39) | 112 (23)

3. Secondary Outcome: Percent Change in Flow Mediated Dilation (FMD)
Description: Endothelial function assessed by flow mediated dilation (FMD). Brachial artery FMD was assessed following overnight fasting. Longitudinal B-mode ultrasound images of the brachial artery, 4-6 cm proximal to the antecubital crease, were obtained using an Aeuson (Mountain View, California) Aspen ultrasoundplatformwith an 11MHZ linear array transducer. lmages were obtained after 10 min of supine relaxation and during reactive hyperemia, induced following in ation of a forearm pneumatic occlusion cuff to supra-systolic pressure (~200 mmHg) for 5 minutes. FMD was defined as the maximum percent change inarterial diameter relative to restingbaseline from 10-120 sec post-deflation of the occlusion cuff.
Time Frame: Baseline, 16 weeks
Population: All completed subjects plus 1 subject in the sertraline arm who did not complete but provided assessment data.
Measure: Number; unit: percentage change
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Number analyzed (Participants) | 36 | 37 | 23
percentage change | 0.2 | 0.9 | 0

4. Secondary Outcome: C-reactive Protein (CRP)
Time Frame: Baseline, 16 weeks
Population: All completed subjects plus 1 subject in the sertraline arm who did not complete but provided assessment data.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Number analyzed (Participants) | 36 | 37 | 23
ug/ml
  Baseline | 2.5 (34) | 2.5 (38) | 2.4 (23)
  16 Week | 2.1 (34) | 2.5 (38) | 2.5 (23)

5. Secondary Outcome: Platelet Factor 4
Time Frame: Baseline, 16 weeks
Population: All completed subjects plus 1 subject in the sertraline arm who did not complete but provided assessment data.
Measure: Mean (Standard Deviation); unit: IU/ml
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Number analyzed (Participants) | 36 | 37 | 23
IU/ml
  Baseline | 44.1 (36) | 34.1 (38) | 32.0 (23)
  16 Week | 35.5 (36) | 34.0 (38) | 34.4 (23)

6. Secondary Outcome: Baroreflex Sensitivity (BRS)
Time Frame: Baseline, 16 weeks
Population: Analysis based on 92 participants with valid baseline measurement.
Measure: Mean (Standard Deviation); unit: msec/mmHg
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Number analyzed (Participants) | 32 | 38 | 22
msec/mmHg
  Baseline | 4.8 (32) | 4.7 (35) | 4.9 (23)
  Week 16 | 4.0 (30) | 5.1 (33) | 4.1 (21)

7. Secondary Outcome: Interleuken 6 (IL-6)
Time Frame: Baseline, 16 weeks
Population: All completed subjects plus 1 subject in the sertraline arm who did not complete but provided assessment data.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Number analyzed (Participants) | 36 | 37 | 23
pg/ml
  Baseline | 1.98 (34) | 1.7 (38) | 1.95 (23)
  16 Week | 1.80 (34) | 2.1 (38) | 1.85 (23)

ADVERSE EVENTS:
Arm/Group | Supervised Aerobic Exercise | Sertraline (Zoloft) | Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/40 | 0/24
Other Adverse Events (participants affected / at risk) | 0/37 | 0/40 | 0/24

LIMITATIONS AND CAVEATS:
Relatively small sample size. Participants had to be willing to accept the condition to which they were randomly assigned, and patients who were not interested in exercise or taking an antidepressant were unlikely to have volunteered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes